CLINICAL TRIAL: NCT04387279
Title: The Effect of Patient's Perceptions for COVID-19 on the Inflammatory Bowel Disease-related Healthcare Utilization in the Hyperepidemic Area
Brief Title: The Impact of COVID-19 on the Health Care Utilization of Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, YooJin Lee, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2020-04-070
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Perception, Self; Facilities and Services Utilization
MeSH Terms: conditions — COVID-19 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inflammatory bowel disease: Patients with inflammatory bowel disease who live in COVID-19 hyperemic area
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Surveys on medical use patterns and patient's perceptions about COVID-19

SUMMARY:
The rapid spread of COVID-19 is expected to have a significant impact on medicine as well as all sectors worldwide. In particular, inflammatory bowel disease (IBD) is a chronic immune disease in which remission and activation are repeated and must be treated consistently throughout life. In addition, patients with IBD may be vulnerable to various infectious diseases due to the immuno-compromised state due to the use of immuno-suppressants or biological agents. During a pandemic, patients with IBD may postpone hospital visits due to concerns about infection with COVID-19, and if they cannot continue drug treatment, there is a concern about the flare up IBD disease activity. Therefore, in this study, we would like to investigate the current status of hospital utilization of IBD patients in Daegu, the epidemic area of COVID-19, and to investigate the effect of patient perception of COVID-19 on hospital ultilization.

DETAILED DESCRIPTION:
Background: In the epidemic area of COVID-19, emergency treatment of chronic diseases other than COVID-19 can be limited. Therefore, it is important to reduce the risk of exposure to COVID-19 in patients with chronic immune diseases such as IBD, but it is most important to manage well so that the underlying diseases are not exacerbated at times when emergency medical treatment may be difficult. However, there is a lack of evidence on the management policy of chronic immune diseases in the current epidemic, and only expert opinions are being presented.

Aim: To investigate the current status of hospital utilization of IBD patients in Daegu, the epidemic area of COVID-19, and to investigate the effect of patient perception of COVID-19 on hospital utilization.

Material and method: This study is a multicenter, prospective, cross-sectional survey which will be consulted in Keimyung University Dongsan Medical Center and Yeungnam University Hospital. Patients with IBD aged above 18 will enrolled and surveyed about their perception about COVID-19 and status of hospital utilization during pandemic period. Patients' demographics and disease-related variables will be evaluated to identify clinical significances.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory growth disease, those who agreed to participate in this study

Exclusion Criteria:

* Those who are unable to understand or answer the questionnaire
* Those who declined to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population will comprise the sample of all patients with inflammatory bowel disease, living in the Daegu city
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Patient's perception of COVID-19 and medical use patterns | 1day
  Correlation between patient's perception of COVID-19 and medical use patterns during the pandemic period

SECONDARY OUTCOMES:
Exacerbation of symptoms | 1day
  Exacerbation of symptoms in patients with IBD during the pandemic period

CONTACTS AND LOCATIONS:
Overall Officials: Yoojin Lee, M.D., Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- KeimyungUniversity, Daegu, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No